CLINICAL TRIAL: NCT04314726
Title: Usefulness of Amelogenins in the Treatment of Periodontal Defects on the Distal Surface of the Lower Second Molar After Adjacent Third Molar Extraction: a Pilot Study
Brief Title: Verify if Amelogenins Had Some Benefits in Improving Lower 2nd Molar Periodontal Healing After 3rd Molar Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Pippi Roberto, MDDS, associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3522/13.02.2015
Record Dates: First submitted 2020-03-10; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Attachment Loss, Periodontal; Teeth, Impacted
Keywords: third molar surgery; amelogenin; periodontal pocket
MeSH Terms: conditions — Periodontal Attachment Loss; Tooth, Impacted; Periodontal Pocket | interventions — Amelogenin

STUDY DESIGN:
Intervention Model Description: A randomized, split-mouth, placebo-controlled, single blind clinical trial, a pilot study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- amelogenins group (Active Comparator): The study involved enrolling 5 periodontitis free patients, to which the extraction of both lower third molars was prescribed. A bone defect at the distal surface of the second molar ≥ 5 mm, had to be present on the intraoral periapical radiography, bilaterally. Amelogenins effect was evaluated by applying them only in the test site and comparing healing results with those obtained on the contra-lateral site
  Interventions: Drug: Amelogenin
- placebo group (Placebo Comparator): The study involved enrolling 5 periodontitis free patients, to which the extraction of both lower third molars was prescribed. A bone defect at the distal surface of the second molar ≥ 5 mm, had to be present on the intraoral periapical radiography, bilaterally. In this group (control site) the conventional treatment was performed, and healing was ensured only by the simple blood clot
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Amelogenin — amelogenins applied on the distal surface of the lower second molar after adjacent third molar extraction
  Other Names: third molar surgery
  Arms: amelogenins group
Drug: Placebos — placebo applied on the distal surface of the lower second molar after adjacent third molar extraction
  Other Names: third molar surgery
  Arms: placebo group

SUMMARY:
Background: Prevention of periodontal defects after the extraction of lower third molars remains a challenge. Various methods have been proposed in the literature, but there are no studies which evaluated the effectiveness of amelogenins.

Methods: A single-blind split-mouth randomized controlled clinical trial (RCT) was performed on 5 patients to verify if amelogenins had some benefits in improving lower second molar periodontal healing after adjacent third molar extraction. A PPD ≥ 8 mm associated with a radiographic bone defect of at least 5 mm were the main inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged < 27, for which the extraction of both lower third molars was indicated
* Bilateral total (bone or osteo-mucosal) third molar impaction
* Bilateral bone defect ≥ 5mm distal to the lower second molars, evaluated on pre- operative periapical radiographs performed with Rinn's film holders
* PPD ≥ 8mm distal to the second lower molars, in at least one of the following probing sites: buccal, disto-buccal, disto-central, disto-lingual
* Intra-operative integrity of both third molar buccal and lingual alveolar cortices

Exclusion Criteria:

* Smoking habit
* Systemic disorders with serious immunologic impairment
* Taking cortisone or other drugs that might interfere with healing process
* Allergy to penicillins
* Previous periodontal treatment
* Less than 2 mm of adherent gingiva at second molar level
* Second molars with a prosthetic crown
* Previous endodontic treatment of second molars
* Furcation involvement of the second molars

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
CAL (Clinical attachment level) pre operative | baseline, pre-surgery
CAL (Clinical attachment level) post operative | 7 days after surgery
CAL (Clinical attachment level) 3 months | 3 months after surgery.
CAL (Clinical attachment level) 12 months | 12 months after surgery.
PPD (Periodontal probing dept) pre operative | baseline, pre-surgery
PPD (Periodontal probing dept) post operative | 7 days after surgery
PPD (Periodontal probing dept) 3 months | 3 months after surgery.
PPD (Periodontal probing dept) 12 months | 12 months after surgery.
REC (recession) pre operative | baseline, pre-surgery
REC (recession) post operative | 7 days after surgery
REC (recession) 3 months | 3 months after surgery.
REC (recession) 12 months | 12 months after surgery.
Radiographic bone Level pre operative | An endoral x-ray was taken baseline, pre-surgery
Radiographic bone Level post operative | An endoral x-ray was taken 7 days after surgery
Radiographic bone Level 3 months | An endoral x-ray was taken 3 months after surgery.
Radiographic bone Level 12 months | An endoral x-ray was taken 12 months after surgery.

SECONDARY OUTCOMES:
Adverse Events pre operative | pre-operative
  the occurrence of adverse events after the use of amelogenins.
Adverse Events post operative | 7 days after surgery
  the occurrence of adverse events after the use of amelogenins.
Adverse Events 3 months | 3 months after surgery.
  the occurrence of adverse events after the use of amelogenins.
Adverse Events 12 months | 12 months after surgery.
  the occurrence of adverse events after the use of amelogenins.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pippi, MDDS, Principal Investigator — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: No